CLINICAL TRIAL: NCT00762619
Title: Clinical Study to Examine Brushing on Dental Implants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Willaim DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRO-2007-IMPLANT-PS
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - (Placebo Comparator): fluoride toothpaste (Ultrabrite)
  Interventions: Drug: Fluoride
- B - Postive control (Active Comparator): fluoride/triclosan/copolymer toothpaste
  Interventions: Drug: Triclosan, fluoride

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Other Names: Ultrabrite toothpaste
  Arms: A -
Drug: Triclosan, fluoride — Brush twice daily
  Other Names: Total toothpaste
  Arms: B - Postive control

SUMMARY:
The efficacy of two dentifrices in controlling gingivitis and plaque in adults with implants

ELIGIBILITY:
Inclusion Criteria:

* Males and females in good oral and general health aged 18 to 76 years.
* A willingness to read, understand, and sign the Informed Consent Form after the nature of the study has been fully explained to them. Subject should demonstrate willingness to comply with all study procedures and availability for duration of study.
* Subjects will use the provided test articles and discontinue the use of other dentifrices and mouthrinses for the duration of the study.
* A minimum of 20 natural teeth with facial and lingual scorable surfaces. Teeth that are grossly carious, fully crowned or extensively restored on facial and/or lingual surfaces, orthodontically banded, abutments, or third molars will not be included in the tooth count.
* Adequate oral hygiene and no signs of oral neglect.
* Subjects will have at least one dental implant and a contralateral natural tooth.
* At the first visit subjects will be examined by a dentist for periodontal health.
* Selected subjects will have periodontal pockets less than 6mm.
* Subjects with gingival index equal to or greater than 1.0 and plaque index equal to or greater than or 1. 5 on the implant tooth will be enrolled. Gingival and plaque indices will be measured during the first visit for the implant. Similarly, these clinical indices (Gingival and plaque index) will be determined for the contralateral natural tooth. (The adjacent teeth will serve as a backup for the studies if control tooth is lost during study).
* Subjects who are habitual users of Colgate Total or other oral hygiene formulations with antimicrobial agents will complete a washout phase of 30 days with a commercial fluoride dentifrice prior to enrollment in the study. This washout dentifrice will be identified and obtained by the clinical investigator from an appropriate local source.

Exclusion Criteria:

* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. Allergy to personal care/consumer products or their ingredients.
* Regular use of mouthwash with antimicrobial agents within the past month.
* History of diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases, e.g. heart disease or AIDS.
* History of hepatitis, rheumatic fever, pacemaker, or prosthetic heart valves, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* Subjects presenting significant medical conditions or need for long term drug therapy.
* Subjects on antibiotic, anti inflammatory or anticoagulant therapy during the month preceding the baseline exam.
* Significant oral soft tissue pathology, systemically related gingival enlargement, severe gingivitis (based on a visual examinations) that would interfere with the study.
* History of active severe periodontal disease with bleeding gums and loose teeth.
* Widespread caries or chronic neglect. Subjects presenting with gross dental caries, severe generalized cervical abrasion and/or enamel abrasion, and large fractured or temporary restorations (based on visual examinations).
* Fixed or removable orthodontic appliance or removable partial dentures.
* Participation in any clinical study including dental plaque/gingivitis clinical trial involving oral care products, within the last 30 days. History of dental prophylaxis or treatments in the month preceding the start of study.
* Self reported pregnancy or lactation.
* History or current use of objects to pierce the lips or tongue.
* Subjects known to be an alcoholic, or a recovering alcoholic.
* History or current use of recreational drugs or narcotics.
* Determine smoking status of subjects and exclude current smokers.
* Determine reason for placing implants in subject to exclude subjects whose implants were placed for trauma.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Mann, MSc, Principal Investigator; Joseph J Zambon, DDS, Principal Investigator
Locations (2):
- State University of New York at Buffalo, Buffalo, New York, United States
- The Hebrew University-Hadassah, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: subjects were screened for medical and oral health criteria and given the assigned study treatment to brush with for the next 6 months. Enrolled subjects all had 1 dental implant and 1 natural tooth identified and used for clinical data information.
Groups:
- A - Fluoride Control: Fluoride toothpaste (Ultrabrite)group contained both 1 natural tooth site and 1 dental implant site for clinical assessment.
- B - Postive Control: fluoride/triclosan/copolymer toothpaste group contained both 1 natural tooth site and 1 dental implant site for clinical assessment.
Period: Overall Study
Arm/Group | A - Fluoride Control | B - Postive Control
Started | 55 | 50
Completed | 55 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Fluoride Control | B - Postive Control | Total
Number analyzed (Participants) | 55 | 50 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 48 | 101
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 54.71 (9.6) | 55.22 (11.6) | 54.95 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 26 | 26 | 52
Region of Enrollment [Number; unit: participants]
  Israel | 55 | 50 | 105

OUTCOME MEASURES:

1. Primary Outcome: Mombelli Plaque Index (mPI) for Natural Teeth
Description: Modified Plaque Index (mPI)is a Dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.96 (0.63) | 1.82 (0.62)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Mombelli Plaque Index (mPI) for Natural Teeth
Description: Modified Plaque Index (mPI) is a Dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 2.05 (0.59) | 1.73 (0.68)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

3. Primary Outcome: Mombelli Plaque Index (mPI) for Dental Implants
Description: as for outcome 2
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.62 (0.63) | 1.35 (0.48)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

4. Primary Outcome: Mombelli Plaque Index (mPI) for Dental Implants
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.71 (0.56) | 1.45 (0.53)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

5. Primary Outcome: Löe-Silness Gingival Index Score (GI) - Natural Teeth
Description: Gingivitis score(GI) is defined: 0 = Absence of inflammation,1 = Mild inflammation-slight change in color and little change in texture,2 = Moderate inflammation-moderate glazing,redness,edema & hypertrophy,3 = Severe inflammation-marked redness and hypertrophy tendency for spontaneous bleeding. Each tooth is scored on 6 surfaces:mesio-facial;2)mid-facial;3)disto-facial;4)mesio-lingual;5)mid-lingualand 6)disto-lingual. A whole mouth score = adding all the GI scores & dividing by the total of number of sites scored. 3rd molars and teeth with restorations or crowns will be excluded.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.3 (0.73) | 1.17 (0.61)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

6. Primary Outcome: Löe-Silness Gingival Index Score (GI) - Natural Teeth
Description: Gingivitis score(GI) is defined: 0 = Absence of inflammation,1 = Mild inflammation-slight change in color and little change in texture,2 = Moderate inflammation-moderate glazing,redness,edema & hypertrophy,3 = Severe inflammation-marked redness and hypertrophy tendency for spontaneous bleeding.Each tooth is scored on 6 surfaces:mesio-facial;2)mid-facial;3)disto-facial;4)mesio-lingual;5)mid-lingualand 6)disto-lingual. A whole mouth score = adding all the GI scores & dividing by the total of number of sites scored. 3rd molars and teeth with restorations or crowns will be excluded.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.29 (0.79) | 1.01 (0.8)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

7. Primary Outcome: Löe-Silness Gingival Index Score (GI)- Dental Implants
Description: Gingivitis Score (GI) is defined: 0 = Absence of inflammation,1=Mild inflammation-slight change in color and little change in texture,2 = Moderate inflammation-moderate glazing,redness,edema & hypertrophy,3 = Severe inflammation-marked redness and hypertrophy tendency for spontaneous bleeding. Each tooth is scored on 6 surfaces:mesio-facial;2)mid-facial;3)disto-facial;4)mesio-lingual;5)mid-lingualand 6)disto-lingual. A whole mouth score=adding all the GI scores & dividing by the total of number of sites scored. 3rd molars and teeth with restorations or crowns will be excluded.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.27 (0.67) | 1.12 (0.63)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

8. Primary Outcome: Löe-Silness Gingival Index Score (GI)- Dental Implants
Description: Gingivitis Score (GI) is defined: 0 = Absence of inflammation,1 = Mild inflammation-slight change in color and little change in texture,2 = Moderate inflammation-moderate glazing,redness,edema & hypertrophy,3 = Severe inflammation-marked redness and hypertrophy tendency for spontaneous bleeding. Each tooth is scored on 6 surfaces:mesio-facial;2)mid-facial;3)disto-facial;4)mesio-lingual;5)mid-lingualand 6)disto-lingual. A whole mouth score=adding all the GI scores & dividing by the total of number of sites scored. 3rd molars and teeth with restorations or crowns will be excluded.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
units on a scale | 1.24 (0.81) | 0.99 (0.73)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

9. Primary Outcome: Gingival Bleeding on Probing (BOP) Using Sulcus Bleeding Index for Teeth
Description: Sulcus bleeding index for teeth is explained here. Gums around teeth are scored:0 = gingiva of normal texture & color, no bleeding;1 = gingiva normal, bleeds on probing;2 = bleeding on probing,change in color, no oedema; 3 = bleeding on probing,change in color, slight oedema;4 = bleeding on probing, change in color, obvious oedema;5=bleeding on probing, spontaneous bleeding, change in color, marked oedema.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
Units on a scale | 0.77 (0.8) | 0.51 (0.67)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

10. Primary Outcome: Gingival Bleeding on Probing (BOP) Using Sulcus Bleeding Index for Teeth
Description: Sulcus bleeding index for teeth is explained here. Gums around teeth are scored:0 = gingiva of normal texture & color, no bleeding;1 = gingiva normal, bleeds on probing;2 = bleeding on probing,change in color, no oedema;3 = bleeding on probing,change in color, slight oedema;4 = bleeding on probing,change in color, obvious oedema;5 = bleeding on probing, spontaneous bleeding,change in color,marked oedema.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
Units on a scale | 0.877 (0.88) | 0.53 (0.76)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

11. Primary Outcome: Gingival Bleeding on Probing (BOP) Using the Modified Sulcus Bleeding Index for Implants
Description: Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
Units on a scale | 0.65 (0.78) | 0.48 (0.68)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

12. Primary Outcome: Gingival Bleeding on Probing (BOP) Using the Modified Sulcus Bleeding Index for Implants
Description: as for outcome 11
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A - Fluoride Control | B - Postive Control
Number analyzed (Participants) | 55 | 50
Units on a scale | 0.81 (0.9) | 0.45 (0.69)
Statistical Analysis 1: Comparison: A - Fluoride Control vs B - Postive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

13. Primary Outcome: A.Actinomycetemcomitans (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are Least means square (LSM)determined by baseline adjusted means including Standard Error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (Colony Forming Units)
Groups:
- A - Fluoride Only Control: Fluoride only (Ultrabrite)
- B - Positive Control: fluoride/triclosan/copolymer toothpaste
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (Colony Forming Units) | 6.269 (0.006) | 5.002 (0.1117)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

14. Primary Outcome: A.Actinomycetemcomitans (DNA Probe Analysis)- Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data point is Least means square (LSM) determined by baseline adjusted means including Standard Error of Means (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.201 (0.1117) | 4.669 (0.1325)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

15. Primary Outcome: A.Actinomycetemcomitans (DNA Probe Analysis)- Dental Implant
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implant. Data point is Least means square (LSM) determined by baseline adjusted means including Standard Error of Means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.814 (0.1262) | 4.446 (0.1589)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

16. Primary Outcome: A.Actinomycetemcomitans (DNA Probe Analysis)- Dental Implant
Description: as for outcome 15
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.664 (0.1222) | 4.339 (0.1908)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

17. Primary Outcome: C.Rectus (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) determined by baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.69 (0.1269) | 3.322 (0.1548)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

18. Primary Outcome: C.Rectus (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 17
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.578 (0.1403) | 2.798 (0.172)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

19. Primary Outcome: C.Rectus (DNA Probe Analysis) - Dental Implant
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) determined by baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.46 (0.1226) | 3.015 (0.1843)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

20. Primary Outcome: C.Rectus (DNA Probe Analysis) - Dental Implant
Description: as for outcome 19
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.318 (0.1318) | 2.758 (0.2106)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

21. Primary Outcome: Capnocytophaga sp. (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 17
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.676 (0.05921) | 4.526 (0.06476)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

22. Primary Outcome: Capnocytophaga sp. (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 17
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.644 (0.07209) | 4.411 (0.07971)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

23. Primary Outcome: Capnocytophaga sp. (DNA Probe Analysis) - Dental Implant
Description: as for outcome 19
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.391 (0.07532) | 4.243 (0.08163)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

24. Primary Outcome: Capnocytophaga sp. (DNA Probe Analysis) - Dental Implant
Description: as for outcome 19
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.356 (0.07716) | 4.268 (0.08752)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

25. Primary Outcome: E.Corrodens (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 13
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.47 (0.1477) | 5.822 (0.1583)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

26. Primary Outcome: E.Corrodens (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 13
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.417 (0.1808) | 5.682 (0.1937)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

27. Primary Outcome: E.Corrodens (DNA Probe Analysis) - Dental Implant
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM)determined by baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.21 (0.148) | 5.639 (0.162)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

28. Primary Outcome: E.Corrodens (DNA Probe Analysis) - Dental Implant
Description: as for outcome 27
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.242 (0.1619) | 5.482 (0.1791)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

29. Primary Outcome: E.Saburreum (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.229 (0.1199) | 4.385 (0.1328)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

30. Primary Outcome: E.Saburreum (DNA Probe Analysis)- Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM)detemined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.079 (0.1424) | 3.571 (0.1655)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

31. Primary Outcome: E.Saburreum (DNA Probe Analysis) - Dental Implant
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.012 (0.1065) | 3.861 (0.1222)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

32. Primary Outcome: E.Saburreum (DNA Probe Analysis) - Dental Implant
Description: as for outcome 31
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.733 (0.1287) | 3.372 (0.1728)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

33. Primary Outcome: F.Nucleatum (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM)determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.337 (0.1773) | 4.403 (0.123)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

34. Primary Outcome: F.Nucleatum (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) detemined by using baseline adjusted means including standard error of means (SEM)
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.243 (0.1265) | 3.405 (0.1327)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

35. Primary Outcome: F.Nucleatum (DNA Probe Analysis) - Dental Implants
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM)determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.89 (0.1277) | 3.637 (0.1354)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

36. Primary Outcome: F.Nucleatum (DNA Probe Analysis) - Dental Implants
Description: as for outcome 35
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.602 (0.1348) | 2.425 (0.1474)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

37. Primary Outcome: Neissera sp. (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.638 (0.1203) | 4.508 (0.1336)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

38. Primary Outcome: Neissera sp. (DNA Probe Analysis) Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points least means square (LSM) determined by baseline adjusted means including standard error of means (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.702 (0.1301) | 4.658 (0.1604)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

39. Primary Outcome: Neissera sp. (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.405 (0.1151) | 3.955 (0.1193)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

40. Primary Outcome: Neissera sp. (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.585 (0.1546) | 4.415 (0.2199)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

41. Primary Outcome: P.Gingivalis (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 34
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.166 (0.1438) | 5.183 (0.1705)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

42. Primary Outcome: P.Gingivalis (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.071 (0.1675) | 4.951 (0.2125)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

43. Primary Outcome: P.Gingivalis (DNA Probe Analysis) - Dental Implants
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) detemined by using baseline adjusted means including standard error of means (SEM)
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.784 (0.1533) | 4.926 (0.1789)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

44. Primary Outcome: P.Gingivalis (DNA Probe Analysis) - Dental Implants
Description: as for outcome 43
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.562 (0.1995) | 4.642 (0.2578)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

45. Primary Outcome: P.Intermedia (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.091 (0.1526) | 3.853 (0.1824)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

46. Primary Outcome: P.Intermedia (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.007 (0.1499) | 3.803 (0.1875)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

47. Primary Outcome: P.Intermedia (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.544 (0.1555) | 3.853 (0.2115)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

48. Primary Outcome: P.Intermedia (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.329 (0.1617) | 3.803 (0.3178)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

49. Primary Outcome: P.Melaninogenica (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.066 (0.1067) | 3.935 (0.1171)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

50. Primary Outcome: P.Melaninogenica (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for both natural teeth. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.062 (0.1141) | 3.691 (0.1252)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

51. Primary Outcome: P.Melaninogenica (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.406 (0.0982) | 3.363 (0.11309)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

52. Primary Outcome: P.Melaninogenica (DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.387 (0.1131) | 3.155 (0.1303)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

53. Primary Outcome: Solobacterium (S.Moorei)(DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.511 (0.1553) | 5.237 (0.1608)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

54. Primary Outcome: Solobacterium (S.Moorei)(DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) determined by using baseline adjusted means including standard error (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.081 (0.2425) | 4.487 (0.2476)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

55. Primary Outcome: Solobacterium (S.Moorei)(DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.767 (0.0346) | 4.701 (0.02777)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

56. Primary Outcome: Solobacterium (S.Moorei)(DNA Probe Analysis) - Dental Implants
Description: as for outcome 31
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.046 (0.3545) | 3.899 (0.4863)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

57. Primary Outcome: Streptococci (DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means )SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.995 (0.1175) | 4.495 (0.1234)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

58. Primary Outcome: Streptococci (DNA Probe Analysis) - Natural Teeth
Description: as for outcome 29
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.867 (0.1195) | 4.109 (0.1255)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

59. Primary Outcome: Streptococci (DNA Probe Analysis) - Dental Implants
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means )SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5 (0.1317) | 3.263 (0.1383)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

60. Primary Outcome: Streptococci (DNA Probe Analysis) - Dental Implants
Description: as for outcome 59
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 4.665 (0.1431) | 2.404 (0.1503)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

61. Primary Outcome: T.Forsythia (DNA Probe Analysis)- Natural Teeth
Description: as for outcome 50
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.408 (0.1348) | 5.143 (0.1474)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

62. Primary Outcome: T.Forsythia (DNA Probe Analysis)-Natural Teeth
Description: as for outcome 29
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.286 (0.1628) | 4.926 (0.182)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

63. Primary Outcome: T.Forsythia (DNA Probe Analysis)- Dental Implants
Description: 14 microorganisms were identified via DNA probe analysis for both Dental Implants. Data points are least means square (LSM) determined by using baseline adjusted means including standard error of means (SEM).
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.19 (0.1637) | 4.628 (0.1831)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

64. Primary Outcome: T.Forsythia (DNA Probe Analysis)- Dental Implants
Description: as for outcome 63
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 6.08 (0.1691) | 4.633 (0.2153)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

65. Primary Outcome: Veillonella sp.(DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) detemined by using baseline adjusted means including standard error (SEM)
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.82 (0.1185) | 4.927 (0.1245)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

66. Primary Outcome: Veillonella sp.(DNA Probe Analysis) - Natural Teeth
Description: 14 microorganisms were identified via DNA probe analysis for natural teeth. Data points are least means square (LSM) determined by using baseline adjusted means including standard error (SEM).
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.746 (0.1282) | 4.563 (0.1346)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

67. Primary Outcome: Veillonella sp.(DNA Probe Analysis) - Dental Implants
Description: 14 microorganisms were identified via DNA probe analysis for Dental Implants. Data points are least means square (LSM) detemined by using baseline adjusted means including standard error (SEM)
Time Frame: 3 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.472 (0.1408) | 4.485 (0.1494)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

68. Primary Outcome: Veillonella sp.(DNA Probe Analysis) - Dental Implants
Description: as for outcome 67
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Log cfu (colony forming units)
Arm/Group | A - Fluoride Only Control | B - Positive Control
Number analyzed (Participants) | 55 | 50
Log cfu (colony forming units) | 5.364 (0.1425) | 4.186 (0.1511)
Statistical Analysis 1: Comparison: A - Fluoride Only Control vs B - Positive Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | A - Fluoride Control | B - Postive Control
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/50
Other Adverse Events (participants affected / at risk) | 0/55 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less